CLINICAL TRIAL: NCT06980545
Title: Phase 3 Study to Evaluate the Role of Total Neoadjuvant Chemotherapy in Partial Responders of Locally Advanced Ovarian Cancer Cancers (NeoPAR Study)
Brief Title: Total Neoadjuvant 6 Cycles of Chemotherapy Versus 3 Cycles in Partial Responder Patients Diagnosed With Epithelial Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed gamal hussein, Assistant lecturer, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoPAR study
Record Dates: First submitted 2025-03-15; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Stage III and IV Ovarian Cancer
MeSH Terms: interventions — Neoadjuvant Therapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- total neoadjuvant 6 cycles of chemotherapy (Experimental): patients who have stationary disease or partial response by MRI after 3 cycles, investigators will give another 3 cycles of chemotherapy to complete six cycles
  Interventions: Drug: Neoadjuvant chemotherapy (Paclitaxel and Carboplatin)

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy (Paclitaxel and Carboplatin) — Neoadjuvant chemotherapy (Paclitaxel and Carboplatin) will be given in complete six cycles

SUMMARY:
neoadjuvant chemotherapy in stage III and IV ovarian cancer is given in 3-4 cycles with patients who R0 surgical resection is less likely to occur, in this study will assess total neoadjuvant chemotherapy 6 cycles then interval debulking surgery (experimental arm) versus 4 cycles then interval debulking surgery (control arm) in patients who achieve partial response or stationary disease by imaging after 3- 4 cycles of neoadjuvant chemotherapy, investigators'' primary end points will be event free survival, safety and tolerability and time to relapse, our secondary end points will be overall survival and surgical morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Recently diagnosed with stage III and IV OC
3. Patients eligible for Platinum-based CTH
4. Patients have PR or SD after 3-4 cycles of NACT

Exclusion Criteria:

1. Relapsed ovarian cancer
2. patients ineligible for Platinum-based CTH
3. Patient not candidate for IDS
4. stage I, II OC
5. Patients progressed after 3 cycles

7-Patients do not tolerate CTH

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
event free survival | it will be measured after 24 months, 36 months and 50 months from neoadjuvant chemotherapy and surgery
  the length of time after primary treatment for a cancer ends that the patient remains free of certain complications or events that the treatment was intended to prevent or delay.
  it will be measured after 24 months, 36 months and 50 months from neoadjuvant chemotherapy and surgery

IPD SHARING:
Plan to Share IPD: Yes